CLINICAL TRIAL: NCT03482817
Title: Drug Cocktail Interaction Study to Investigate the Effect of St. John's Wort Dry Extract Ze 117 on Several Cytochrome P450 Enzymes and on Transporter P-Glycoprotein in Healthy Volunteers
Brief Title: Drug Cocktail Interaction Study of St. John's Wort Dry Extract Ze 117
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Max Zeller Soehne AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ze117-1-2017-01
Record Dates: First submitted 2018-02-26; First posted 2018-03-29 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Drug Interaction Study
MeSH Terms: interventions — ZE 117

STUDY DESIGN:
Intervention Model Description: open-label, non-randomized, single-sequence study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Probe drug cocktail / Ze 117 (Experimental): One-sequence, Probe drug cocktail alone and in combination with Ze 117.
  Interventions: Drug: Ze 117; Drug: Probe drug cocktail

INTERVENTIONS:
Drug: Ze 117 — Subjects will be hospitalized to receive a probe drug cocktail alone and in combination with Ze 117.
  Other Names: St. John's wort dry extract Ze 117
Drug: Probe drug cocktail — Subjects will be hospitalized to receive a probe drug cocktail alone and in combination with Ze 117.

SUMMARY:
This Study evaluates the Effect of St. John's Wort dry Extract Ze 117 on Several Cytochrome P450 Enzymes and on Transporter P-Glycoprotein in Healthy Volunteers.

DETAILED DESCRIPTION:
Current data indicate that St. John's wort preparations may induce hepatic cytochrome P450 enzymes and transport proteins. This can result in drug interactions.

The study design is standard for DDI studies and is based on the regulatory guidance of the Food and Drug Administration (FDA) and of the European Medicines Agency (EMA).

A cocktail approach involving the administration of multiple cytochrome P450 (CYP)- or P-glycoprotein (P-gp)-specific probe drugs is used to simultaneously assess the activities of these enzymes and the transporter P-gp.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* Caucasian male or female subjects aged between ≥18 and ≤55years
* Physically and mentally healthy
* BMI between ≥19 and ≤29 kg/m2, and body weight ≤90 kg
* Non-smoker
* If female, the pregnancy test at screening and at admission must be negative

Exclusion Criteria:

* Known or suspected hypersensitivity to study drugs
* history of, any clinically significant diseases
* Positive test of hepatitis B, hepatitis C or HIV Screening
* Known photohypersensitivity

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Caucasian
Enrollment: 20 (Estimated)
Dates: Start 2018-02-05 (Actual); Primary Completion 2018-05-17 (Estimated); Study Completion 2018-06-23 (Estimated)

PRIMARY OUTCOMES:
Area under the Plasma concentration versus time curve (AUC0-t) | 72 hours
  Pharmacokinetic Parameter AUC0-t (mg*h/L) of the probe drugs will be determined.

SECONDARY OUTCOMES:
Area under the Plasma concentration versus time curve (AUC0-inf) | 72 hours
  Pharmacokinetic parameter (mg*h/L) of the probe drugs and their metabolites will be determined.
Peak Plasma Concentration (Cmax) | 72 hours
  Pharmacokinetic Parameter (ng/ml) of the probe drugs and their metabolites will be determined.
Elimination rate constant (Ke) | 72 hours
  Pharmacokinetic Parameter (h^-1) of the probe drugs and their metabolites will be determined.
Elimination half life (t1/2) | 72 hours
  Pharmacokinetic Parameter (h) of the probe drugs and their metabolites will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lissy, Principal Investigator — Neu-Ulm
Locations (1):
- Nuvisan GmbH, Neu-Ulm, Germany

IPD SHARING:
Plan to Share IPD: Undecided